CLINICAL TRIAL: NCT05694221
Title: A Single-centre, Open Labeled, Fixed-sequence Study to Evaluate the Effect of Supaglutide on Digoxin or Metformin Pharmacokinetics
Brief Title: Drug Drug Interaction (DDI) Between Supaglutide and Digoxin or Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: YN011-D01
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Digoxin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Digoxin combined with Supaglutide group (Experimental): Subjects will receive a single oral dose of 0.25 mg digoxin tablets on Day 1. And will received subcutaneous injection of sulpalutide QW for five weeks（D5-D33）.
  Then receive another single oral dose of 0.25 mg digoxin tablets on Day 35.
  Interventions: Drug: Supaglutide injection; Drug: Digoxin
- Group B: Metformin combined with Supaglutide Group (Experimental): Subjects will receive multiple oral dose of Metformin tablets on Day 1-3. And will received subcutaneous injection of sulpalutide QW for five weeks（D5-D33）.
  Then receive another round of Metformin tablets on Day 32-34.
  Interventions: Drug: Supaglutide injection; Drug: Metformin

INTERVENTIONS:
Drug: Supaglutide injection — Administered subcutaneously in the Supaglutide arms
  Other Names: Diabegone
Drug: Digoxin — Oral Administration
  Other Names: Digoxin Tablets
  Arms: Group A: Digoxin combined with Supaglutide group
Drug: Metformin — Oral Administration
  Other Names: Glucophage
  Arms: Group B: Metformin combined with Supaglutide Group

SUMMARY:
This is a study of a drug drug interaction between Supaglutide and Digoxin or Metformin.

DETAILED DESCRIPTION:
This is a single-centre, open labeled, fixed-sequence study designed to assess the pharmacokinetic effects of multiple subcutaneous injections of Supalutide on a single oral dose of digoxin or multiple oral doses of metformin. 32 healthy subjects are planned to be enrolled and allocated to 2 parallel trial groups, Digoxin combined with Sulpalutide injection (Group A) and Metformin combined with Sulpalutide injection (Group B), with 16 cases in each group, of which no less than 4 were of a single sex.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese subjects.
2. Age between 18 and 45 years, inclusive.
3. Body mass index [BMI = weight (kg)/height2 (m2)] of between 20 and 28 kg/m2 (including thresholds), with male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg.
4. Subjects with no plan of pragnancy within the screening period up to 3 months after the last dose and who are voluntarily using contraception.

6. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Subjects with a previous or existing history of serious cardiac, hepatic, renal, gastrointestinal, neurological, psychiatric abnormalities and metabolic abnormalities.
2. Subjects with a previous or existing disease affecting the absorption, distribution, metabolism or excretion of drugs, such as active peptic ulcers or bleeding, history of ulcers or bleeding, acute and chronic pancreatitis, etc.
3. Subjects with a history or family history of C-cell tumours/carcinoma of the thyroid gland, or a previous history of thyroid insufficiency or thyroid hormone abnormalities
4. Subjects who have undergone major surgery within 4 weeks prior to screening which, in the judgment of the investigator, may affect this trial, such as gastric and duodenal surgery, cholecystectomy, nephrectomy, or removal of malignant tumours (except for previous appendectomy), or those who are scheduled to undergo major surgery during the trial
5. those with existing symptoms of unexplained infection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Group A: Plasma Cmax of digoxin | 39 Days
  when given in combination with supaglutide in healthy volunteers
Group A: Plasma AUC0-last of digoxin | 39 Days
  when given in combination with suplaglutide in healthy volunteers
Group A: Plasma AUC0-inf of digoxin | 39 Days
  when given in combination with supaglutide in healthy volunteers
Group B: Plasma Cmax,ss of Metformin | 34 Days
  when given in combination with supaglutide in healthy volunteers
Group B: Plasma AUC0-tau of Metformin | 34 Days
  when given in combination with suplaglutide in healthy volunteers

SECONDARY OUTCOMES:
Group A: Plasma Tmax of Digoxin | 39 Days
  when given in combination with supaglutide in healthy volunteers
Group A: Plasma t1/2 of digoxin | 39 Days
  when given in combination with supaglutide in healthy volunteers
Group A: Plasma CL/F of digoxin | 39 Days
  when given in combination with suplaglutide in healthy volunteers
Group A: Plasma Vz/F of digoxin | 39 Days
  when given in combination with supaglutide in healthy volunteers
Group B: Plasma Tmax of Metformin | 34 Days
  when given in combination with supaglutide in healthy volunteers
Group B: Plasma Cmin,ss of Metformin | 34 Days
  when given in combination with suplaglutide in healthy volunteers
Group B: Plasma t1/2 of Metformin | 34 Days
  when given in combination with suplaglutide in healthy volunteers
Group B: Plasma CL/F of Metformin | 34 Days
  when given in combination with suplaglutide in healthy volunteers
Group B: Plasma Vz/F of metformin | 34 Days
  when given in combination with suplaglutide in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, He J, Wu J, Liu W, Xu Y, Li Y, Zhang J, Wang Q. Effect of Efsubaglutide Alfa on the Pharmacokinetics of Metformin and Digoxin in Healthy Participants. Clin Pharmacokinet. 2025 Sep;64(9):1367-1377. doi: 10.1007/s40262-025-01541-0. Epub 2025 Jun 30. PMID 40587051